CLINICAL TRIAL: NCT00765661
Title: A Phase 2, Open-Label, Multi-Center, Randomized Trial To Demonstrate The Pharmacokinetics Of LCP-Tacro™ Tablets Once Daily and Prograf® Capsules Twice Daily In Adult De Novo Kidney Transplant Patients
Brief Title: Pharmacokinetics of LCP-Tacro(TM) Once Daily And Prograf® Twice A Day in Adult De Novo Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other); Aptuit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCP - Tacro 2017
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Failure; Renal Failure
Keywords: Kidney; Transplantation; Immunosuppression; Tacrolimus; Prograf
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Experimental): The initial dose starting at 0.14 mg/kg (the starting daily dose for African-American patients was 0.17 mg/kg), will be administered orally in the morning (before noon) within 12 hours after transplantation. Subsequent doses adjusted to maintain a target whole blood tacrolimus trough level of 7 - 20 ng/mL for the remainder of the pharmacokinetic (PK) phase of the study (through Study Day 14). Post PK patient enter the maintenance phase of the study and remain on assigned study drug until Study Day 360. Dose of study drug was adjusted to maintain tacrolimus trough levels between 5 - 20 ng/mL from Day 15 until Day 90 and then between 5 - 15 ng/mL for the remainder of the study according to local standard of care.
  Interventions: Drug: Tacrolimus (Tacro™)
- Prograf (tacrolimus) (Active Comparator): Starting total daily dose of 0.10 mg/kg administered in two equally divided doses, morning and evening, per product labeling. Subsequent doses adjusted to maintain a target whole blood tacrolimus trough level of 7 - 20 ng/mL for the remainder of the pharmacokinetic (PK) phase of the study (through Study Day 14). Post PK patient enter the maintenance phase of the study and remain on assigned study drug until Study Day 360. Dose of study drug was adjusted to maintain tacrolimus trough levels between 5 - 20 ng/mL from Day 15 until Day 90 and then between 5 - 15 ng/mL for the remainder of the study according to local standard of care.
  Other name: tacrolimus
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Tacrolimus (Tacro™) — The initial dose at 0.14 mg/kg (daily dose for African-American is 0.17 mg/kg), oral in the morning (before noon) within 12 hours after transplantation. Subsequent doses adjusted to maintain a target tacrolimus trough level of 7 - 20 ng/mL for (PK) phase of the study (through Study Day 14). Post PK maintenance phase of the study and remain on assigned study drug until Study Day 360. Dose of study drug was adjusted to maintain tacrolimus trough levels between 5 - 20 ng/mL from Day 15 until Day 90 and then between 5 - 15 ng/mL for the remainder of the study according to local standard of care.
  Other Names:
  Tacrolimus modified-release
  Other Names: LCP -Tacro
  Arms: LCP-Tacro
Drug: Prograf — Prograf® capsules, twice daily: Starting total daily dose of 0.10 mg/kg administered in two equally divided doses, morning and evening, per product labeling. Subsequent doses adjusted to maintain a target whole blood tacrolimus trough level of 7 - 20 ng/mL for the remainder of the pharmacokinetic (PK) phase of the study (through Study Day 14). Post PK patient enter the maintenance phase of the study and remain on assigned study drug until Study Day 360. Dose of study drug was adjusted to maintain tacrolimus trough levels between 5 - 20 ng/mL from Day 15 until Day 90 and then between 5 - 15 ng/mL for the remainder of the study according to local standard of care.
  Other name: tacrolimus
  Other Names: tacrolimus
  Arms: Prograf (tacrolimus)

SUMMARY:
The purpose of this study is to demonstrate the pharmacokinetics (PK, measuring the amount of medication in blood samples) and safety of a new medicine, LCP-Tacro™ tablets, and Prograf® capsules, a drug commonly taken by transplant recipients to prevent the body from rejecting a transplanted kidney. LCP-Tacro is a tablet containing the same active ingredient (tacrolimus) that is in Prograf capsules, but the tablet has been designed to release tacrolimus over an extended period so that it only has to be taken once daily. LCP-Tacro is an investigational drug.

This study will evaluate the levels of tacrolimus in the blood in the first two weeks after a kidney transplant in patients randomly assigned (by chance, like flipping a coin) to take either LCP-Tacro™ tablets (tacrolimus) once daily or Prograf® capsules twice daily. In addition, patients will remain on study drug for 360 days in order to evaluate the relative safety of LCP-Tacro™ tablets compared to Prograf over a longer period of time.

DETAILED DESCRIPTION:
This study was a randomized, parallel-group, open label, multicenter study in adult de novo kidney transplant patients to demonstrate the pharmacokinetics and safety of LCP-Tacro tablets and Prograf capsules in the first 2 weeks after kidney transplantation. In addition the study compared the efficacy and safety of LCP-Tacro and Prograf over an additional 50 weeks after kidney transplantation. Eligible patients were randomized (1:1 ratio) within 12 hours after transplantation (Day 0) to receive either: 1) LCP-Tacro tablets orally once daily (QD) in the morning, with an interval of 24+/- hours between doses, starting at 0.14 mg/kg (the starting daily dose for African-American patients was 0.17 mg/kg), or 2) Prograf capsules in 2 equally divided doses for African-American patients was (0.2 mg/kg total daily dose) as recommended in the U.S. Prescribing Information (Astellas Pharma US, April 2006). Day 1 was defined as the day on which the first morning dose of study medication was given which was to be within 48 hours of transplantation. Subsequent doses of study medication were adjusted to maintain target whole blood tacrolimus trough level of 7 to 20 ng/mL for the remainder of the pharmacokinetic phase of the study (Day1 through Day 14). Twenty-four-hour pharmacokinetic assessments were performed on Days 1, 7, and 14. Following completion of the third and final pharmacokinetic assessment on the morning of Day 14, patients entered the maintenance phase (Days 15 to 360) of the study and remained on their assigned study medication until Day 360. Visits for safety assessments and tacrolimus trough levels during the maintenance phase were on Days 42, 90, 120, 180, 270, and 360. On Day 360, the patients were placed on a maintenance immunosuppressive regimen determined by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women at least 18 years of age who are recipients of a kidney transplant from a deceased donor or a live donor and who receive their first oral dose of randomized study drug within 48 hours of the transplant surgery (graft reperfusion)

Exclusion Criteria:

* Recipient of any transplanted organ other than a kidney
* Recipients of a kidney from a non-heart beating donor
* Recipients of a kidney from an ABO incompatible donor
* Recipients of a kidney with a cold ischemia time of ≥ 36 hours
* Recipients of a bone marrow or stem cell transplant
* Patients with a white blood cell count ≤ 2.8 x 109/L unless the absolute neutrophil count (ANC) is > 1.0 x 109/L
* Patients with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) enzyme levels > 3 times the upper limit of normal during the 30 days prior to the transplant procedure
* Patients who fail a drugs of abuse screen
* Patients unable to swallow study medication
* Patients incapable of understanding the purposes and risks of the study, who cannot give written informed consent, or who are unwilling to comply with the study protocol
* Pregnant or nursing women (women of childbearing potential must have a negative serum pregnancy test within seven days prior to receiving study medication)
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception throughout the duration of the study
* Patients who were treated with any other investigational agent in the 30 days prior to enrollment
* Patients who are hepatitis C virus (HCV) negative who have received a HCV positive (HCV RNA by polymerase chain reaction (PCR) or HCV antibody) donor kidney
* Patients seropositive for human immunodeficiency virus (HIV)
* Patients with a current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully
* Patients with uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patients with severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patients with a known hypersensitivity to tacrolimus
* Patients with any form of current substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Alloway, PharmD, Principal Investigator — University of Cincinnati, allowarr@ucmail.uc.edu
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Randomized, parallel group, open-label, multi-center study in adult de novo kidney transplant patients to demonstrate the pharmacokinetics and safety of LCP-Tacro tablets in the first 2 weeks after kidney transplantation. Eligible patients were randomized (1:1 ratio) within 12 hours after transplantation (Day 0) to receive LCP-Tacro tablets orally once daily (QD) in the morning, with an interval of 24 +/-1 hours between doses, starting at 0.14 mg/kg (the starting daily dose for African-American patients was 0.17 mg/kg)
- Group B: Randomized, parallel-group, open-label, multi-center study in adult de novo kidney transplant patients to demonstrate the pharmacokinetics and safety of Prograf capsules in the first 2 weeks after kidney transplantation. Eligible patients were randomized (1:1 ratio) within 12 hours after transplantation (Day 0) to receive Prograf capsules in 2 equally divided doses, starting at 0.1 mg/kg every 12 hours (0.2 mg/kg total daily dose) as recommended in the U.S. Prescribing Information
Period: Overall Study
Arm/Group | Group A | Group B
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gorup A: LCP - Tacro™ tablets, once daily (LifeCycle Pharma A/S, Hørsholm DK)
  tacrolimus (Tacro™): LCP - Tacro™ tablets, orally
- Group B: Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
  Prograf®: Prograf® capsules, twice daily, orally
- Total: Total of all reporting groups
Arm/Group | Gorup A | Group B | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12) | 46.1 (13.87) | 47.7 (12.94)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 31 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 9 | 30
  Male | 11 | 22 | 33
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of LCP-Tacro™ Tablets in the First 14 Days After Transplantation in Adult de Novo Kidney Recipients.
Description: Comparison of the proportion of patients achieving sufficient tacrolimus whole blood trough levels (7 to 20 ng/mL) during the first 14 days post-transplantation
Time Frame: 14 days
Measure: Number; unit: percentage of patients
Groups:
- Group A: LCP - Tacro™ tablets, once daily (LifeCycle Pharma A/S, Hørsholm DK) tacrolimus (Tacro™)
- Group B: Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 28 | 28
percentage of patients | 78.57 | 57.14

2. Secondary Outcome: Comparative Pharmacokinetics Between LCP-Tacro and Prograf Within 14 Days After Kidney Transplantation.
Description: To compare the pharmacokinetics (AUC, Cmax, C24/Cmin) on Days 1, 7 and 14 of LCP-Tacro with the pharmacokinetics of Prograf in adult de novo kidney transplant patients.
Time Frame: 14 days
Population: The outcome measure is listed as arithmetic mean of the pharmacokinetic parameters for raw data (not dose corrected) for tacrolimus in the ITT population on Day 14.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 28 | 28
ng/mL
  Cmax | 28.21 (13.68) | 20.27 (6.49)
  Cmin | 10.37 (4.24) | 8.12 (3.13)

3. Secondary Outcome: Comparative Pharmacokinetics Between LCP-Tacro and Prograf Within 14 Days After Kidney Transplantation.
Description: as for outcome 2
Time Frame: 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 28 | 28
ng*hr/mL | 349.31 (112.41) | 255.22 (80.39)

4. Secondary Outcome: Evaluation of Safety and Efficacy of LCP-Tacro Compared to Prograf in Adult de Novo Kidney Transplant Patients.
Description: To evaluate the efficacy and safety of LCP-Tacro compared to Prograf in the first 12 months after kidney transplantation.
  Efficacy was assessed by monitoring biopsy-proven acute rejection (BPAR) according to the Banff criteria, graft failure (defined by a patient starting dialysis for at least 30 days, nephrectomy, retransplantation, or death with a functioning graft), patient survival, and renal function based on serum creatinine and glomerular filtration rate (GFR), based on serum creatinine, serum urea nitrogen, and serum albumin.
Time Frame: 12 months
Population: All patients receiving at least one dose of study drug was included in the safety evaluation.
Measure: Number; unit: participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 32 | 31
participants
  BPAR | 0 | 0
  Graft Failure | 0 | 2
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 and up to end of study for a total of 12 months.
Groups:
- Group A: LCP - Tacro™ tablets, once daily (LifeCycle Pharma A/S, Hørsholm DK)
  tacrolimus (Tacro™): LCP - Tacro™ tablets
- Group B: Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
  Prograf®: Prograf® capsules, twice daily
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 15/32 | 17/31
Other Adverse Events (participants affected / at risk) | 32/32 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=32) | Group B (N=31)
gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
localized infection (Infections and infestations) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
vomitting (Gastrointestinal disorders) | 1 (2) | 0 (0)
urosepsis (Infections and infestations) | 1 (1) | 0 (0)
acute renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
serum sickness (Immune system disorders) | 0 (0) | 1 (1)
haemturia (Renal and urinary disorders) | 0 (0) | 1 (1)
wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
renal lymphocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
oesphagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
lymphocele (Vascular disorders) | 0 (0) | 1 (1)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
viral infection (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
anemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
coagulophathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
internal normalized ratio increase (Investigations) | 0 (0) | 1 (1)
renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
drug intolerance (General disorders) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=32) | Group B (N=31)
Anaemia (Blood and lymphatic system disorders) | 13 (15) | 14 (19)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 9 (10) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 3 (3)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 6 (7)
Abdominal lower pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (17) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 16 (21) | 17 (21)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (22) | 17 (22)
Vomiting (Gastrointestinal disorders) | 10 (12) | 7 (8)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (5)
Gait disturbance (General disorders) | 1 (1) | 2 (2)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Oedema (General disorders) | 2 (2) | 2 (3)
Oedema peripheral (General disorders) | 9 (9) | 10 (13)
Pyrexia (General disorders) | 5 (5) | 6 (8)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 3 (3)
BK virus infection (Infections and infestations) | 2 (2) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Human papylomavirus infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 6 (7)
Urinary tract infection (Infections and infestations) | 12 (21) | 12 (19)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Drug toxicity (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Prost procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 7 (9) | 6 (7)
Blood creatinine increased (Investigations) | 8 (11) | 7 (8)
Liver function test abnormal (Investigations) | 1 (1) | 3 (4)
Weight increased (Investigations) | 4 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 4 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Fluid overload (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (8) | 10 (13)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (13) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 10 (12) | 7 (7)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 4 (6)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 6 (6) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (5) | 5 (5)
Depression (Psychiatric disorders) | 2 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 11 (13) | 6 (6)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (6) | 5 (7)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (4) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Wound drainage (Surgical and medical procedures) | 2 (2) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 10 (13) | 8 (11)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Lymphocele (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study is a multicenter collaborative investigation and the clinical trial results are to be published as a collaborative manuscript. Authorship will reflect varying levels of individual contribution to the study by the individual PIs.